CLINICAL TRIAL: NCT02869126
Title: Study of the Concordance Between a Traditional Protocol of Stress and Rest Myocardial Tomoscintigraphy Using 99mTc-sestamibi and a Double Isotope Protocol Using Thallium-201 and 99mTc-sestamibi, With a Semiconductor Camera
Brief Title: Stress and Rest Myocardial Tomoscintigraphies Using Mono- or Double-isotope Protocol With a Semiconductor Camera
Acronym: D-SPECT BIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-A00569-34
Record Dates: First submitted 2016-08-09; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Myocardial Perfusion
Keywords: 99mTc-Sestamibi; thallium-201; semiconductor camera
MeSH Terms: interventions — Technetium Tc 99m Sestamibi; Thallium-201

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Experimental): Patients with abnormalities of myocardial perfusion detected with stress tomoscintigraphy, undergo double isotope myocardial tomoscintigraphy using Thallium-201 and 99mTc-sestamibi and traditional myocardial tomoscintigraphy using 99mTc-sestamibi with a semiconductor camera
  Interventions: Procedure: Tomoscintigraphy with D.SPECT camera (SPECTRUM Dynamics®, Israel); Drug: 99mTc-Sestamibi; Drug: Thallium-201

INTERVENTIONS:
Procedure: Tomoscintigraphy with D.SPECT camera (SPECTRUM Dynamics®, Israel) — * During stress test, intravenous injection of 99mTc-Sestamibi (between 80 and 150 MBq according to weight) in patient
  * Stress conventional acquisition with D.SPECT camera 20 min after injection
  * 60 min after 99mTc-Sestamibi injection, rest injection of thallium-201 (50% activity of stress 99mTc-Sestamibi)
  * double isotope acquisition 5 min after thallium-201 injection
  * injection of 99mTc-Sestamibi at rest (activity 3 times higher), after 2 hours from first 99mTc-Sestamibi injection
  * rest conventional acquisition 20 min later
Drug: 99mTc-Sestamibi — First intravenous injection between 80 and 150 MBq according to patient weight and second injection with 3-time-higher activity, 2 hours after the first
  For tomoscintigraphy
Drug: Thallium-201 — Injection of thallium-201 (50% activity of first 99mTc-Sestamibi injection)
  For tomoscintigraphy

SUMMARY:
The purpose is to demonstrate the concordance of diagnostic information obtained with:

1. a conventional examination with 2 distinct recordings on D.SPECT camera after 99mTc-sestamibi injections, the first post-stress and the second at rest, 2 to 3 hours later,

   and
2. a double isotope examination with a supplementary recording after injection of a little activity of thallium-201 at rest after the first recording and before the second injection of 99mTc-sestamibi for conventional recording at rest,

in patients showing abnormalities of myocardial perfusion in stress myocardial tomoscintigraphy.

DETAILED DESCRIPTION:
Myocardial perfusion tomoscintigraphy is very used for diagnosis and characterization of abnormalities of stress and rest myocardial perfusion. This examination can be performed with semiconductor gamma cameras that are more performant than conventional cameras regarding spatial resolution, detection sensitivity and energy resolution.

The amelioration of energy resolution could allow the realization of simultaneous recordings of a dye injected at rest and another injected during stress (double isotope recording), while conventional examination needs 2 different recordings, stress and rest, separated from several hours.

In this study patients undergo a conventional examination with D.SPECT camera with 2 recordings, the first after injection of a little activity of 99mTc-sestamibi at stress (≤ 100 MBq) and the second, 2 hours later, after injection at rest of a 3 time bigger activity of 99mTc-sestamibi (≤ 300 MBq). An activity of thallium-201(≤ 50 MBq) is injected at rest after the first recording of stress. 5 minutes later, a supplementary double isotope recording is realized with D.SPECT camera (99mTc-Sestamibi-stress / thallium201-rest).

The demonstration of the hypothesis of this study could considerably diminish the duration of the examination (from 3 to 4 hours to less than 1 hour).

ELIGIBILITY:
Inclusion Criteria:

* > 18, without guardianship, signed informed consent
* Without contraindication for myocardial perfusion tomoscintigraphy and stress technique (dipyridamole and/or effort), according to common criteria to French Societies of Cardiology and Nuclear Medicine, as it is requested for all patients needing this routine examination
* Not in life-and-death emergency, with a stable clinical state (without cardiac insufficiency or instable coronary, without hypertension not well-stabilized under treatment)
* Effective contraceptive method for women of childbearing potential
* Weight ≤ 100 kg (> 100 kg patients need higher injected activities in order to obtain adequate image quality)
* Perfusion abnormalities on stress images

Exclusion Criteria:

* < 18
* Contraindications to stress test (effort and/or dipyridamole)
* Hypersensibility to thallium201 chloride or one of excipients
* Claustrophobic patient or incapable to stay lying down for 30 minutes
* Pregnancy or doubt of pregnancy
* Breastfeeding woman
* Weight > 100 kg
* Non affiliation to social security plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2012-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Quality of images obtained with double isotope tomoscintigraphy and conventional tomoscintigraphy | day 0
  Bad; medium; good; very good
Nature of observed abnormalities obtained with double isotope tomoscintigraphy and conventional tomoscintigraphy | day 0
  Without abnormalities or artefacts (normal); with rest reversible abnormalities (ischemia); with rest non reversible abnormalities (infarction)

CONTACTS AND LOCATIONS:
Overall Officials: Wassila DJABALLAH, Dr, Principal Investigator — Service de Médecine Nucléaire, Hôpital de Brabois, 54511 Vandœuvre les Nancy
Locations (2):
- France (2):
  - Service de Médecine Nucléaire - CLCC Jean Perrin, Clermont-Ferrand
  - Service de Médecine Nucléaire - Hôpital de Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No